CLINICAL TRIAL: NCT07249502
Title: The Effects of Scoliosis-Specific Corrective Exercises on Physical Fitness Parameters in Adolescents With Idiopathic Scoliosis
Brief Title: Scoliosis-Specific Exercises on Physical Fitness Parameters
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Tuğçe Yavuz, Principal Investigator, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25-119
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Idiopathic Adolescent; Scoliosis Idiopathic Adolescent Treatment
Keywords: Scoliosis; Scoliosis-Specific Corrective Exercises; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scoliosis-Specific Corrective Exercise Group (Experimental): Participants in this group will receive an individualized scoliosis-specific corrective exercise program based on the Schroth classification. The program focuses on three-dimensional spinal correction and stabilization. Each participant will attend supervised sessions delivered by a Schroth-certified physiotherapist for 45-60 minutes, twice per week, for a total of 16 sessions over 8 weeks. Home exercises will also be prescribed and monitored for adherence.
  Interventions: Behavioral: Scoliosis-Specific Corrective Exercise Program
- Postural Education Control Group (Active Comparator): Postural education and basic corrective exercise elements performed at home 2 times per week for 8 weeks.
  Interventions: Behavioral: Postural Education and Basic Corrective Exercises

INTERVENTIONS:
Behavioral: Scoliosis-Specific Corrective Exercise Program — An individualized scoliosis-specific corrective exercise program based on the Schroth method, delivered by a certified physiotherapist twice per week for 8 weeks.
  Arms: Scoliosis-Specific Corrective Exercise Group
Behavioral: Postural Education and Basic Corrective Exercises — Postural education and basic corrective exercise elements to be performed at home twice per week for 8 weeks.
  Arms: Postural Education Control Group

SUMMARY:
Adolescent Idiopathic Scoliosis is a common musculoskeletal condition characterized by a three-dimensional spinal deformity, affecting approximately 2-4% of adolescents worldwide and occurring more frequently in girls. Beyond spinal curvature, Adolescent Idiopathic Scoliosis can negatively influence physical fitness, muscular strength, respiratory function, postural control, and participation in daily activities. These factors may reduce overall functional capacity and quality of life.

Scoliosis-specific corrective exercises, including approaches such as Schroth and The Scientific Exercise Approach to Scoliosis, have been shown to improve postural symmetry, slow curve progression, and enhance respiratory and psychosocial outcomes. However, the effects of these exercises on physical fitness parameters-such as muscle strength, flexibility, motor performance, and cardiorespiratory endurance-remain insufficiently studied.

The aim of this study is to investigate the effects of scoliosis-specific corrective exercises on physical fitness parameters in adolescents diagnosed with Adolescent Idiopathic Scoliosis. Measures of strength, flexibility, motor performance, and cardiorespiratory endurance will be assessed before and after the intervention. Findings from this study are expected to contribute to the development of evidence-based conservative treatment protocols focusing not only on curve progression but also on functional capacity and overall fitness in adolescents with scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Adolescent Idiopathic Scoliosis confirmed by an orthopedic specialist
* Cobb angle between 10° and 45° on standing anteroposterior radiograph
* Age between 10 and 19 years
* No prior history of scoliosis-specific exercise treatment
* Ability to participate regularly in the exercise program -Voluntary willingness to participate in the study -

Exclusion Criteria:

* Presence of mental, rheumatologic, neuromuscular, cardiovascular, or pulmonary disorders
* Pain or orthopedic conditions that prevent participation in exercise
* Visual and/or hearing impairments affecting communication or assessment
* History of spinal surgery, spinal tumor, or related interventions
* Any medical condition for which exercise is contraindicated
* Communication difficulties that limit participation

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-19 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength | 8 weeks
  Muscle strength of the quadriceps, middle deltoid, and handgrip will be assessed using a handheld dynamometer. The change in strength from baseline to 8 weeks will be analyzed.

SECONDARY OUTCOMES:
Aerobic Capacity | 8 weeks
  Aerobic capacity will be assessed using the Six Minute Walk Test. The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. The total meter of completed laps will be recorded, and the change from baseline to 8 weeks will be analyzed.
Sit and Reach Test | 8 weeks
  Flexibility of the lower extremity and trunk will be assessed with the Sit-and-Reach Test. Scores will be recorded in centimeters, and changes from baseline to 8 weeks will be evaluated.
Shoulder Mobility Test | 8 weeks
  Upper extremity flexibility will be assessed using the Shoulder Mobility Test. The distance between fingertips will be recorded as positive or negative values. Changes between baseline and 8 weeks will be analyzed.
Y-Balance Test | 8 weeks
  Dynamic balance performance will be measured using the Y-Balance Test in three directions (anterior, posteromedial, posterolateral). Reach distances will be normalized to leg length. Change from baseline to 8 weeks will be evaluated.
Body mass index | 8 weeks
  Body mass index will be calculated to assess general adiposity. Body mass index will be computed as weight (kg) divided by height squared (m²). Participants will be classified according to World Health Organization (WHO) Body mass index categories.
waist circumference | 8 weeks
  Waist circumference will be measured to evaluate central (abdominal) adiposity. Measurements will be taken using a non-elastic tape measure placed horizontally at the midpoint between the lowest rib and the iliac crest. Participants will stand upright with feet shoulder-width apart and arms relaxed. The measurement will be recorded at the end of a normal expiration to the nearest 0.1 cm.
Hip Circumference waist circumference | 8 weeks
  Hip circumference will be measured to assess gluteofemoral adiposity. A non-elastic tape measure will be placed horizontally around the widest part of the buttocks, ensuring the tape remains parallel to the floor. Participants will stand in a relaxed position, and the measurement will be recorded to the nearest 0.1 cm without compressing the skin.
Neck Circumference | 8 weeks
  Neck circumference will be measured as an indicator of upper-body adiposity. Using a flexible, non-stretch tape, the circumference will be taken at the level just below the laryngeal prominence (Adam's apple) while the participant stands upright and looks straight ahead. The tape will be positioned perpendicular to the long axis of the neck, and measurements will be recorded to the nearest 0.1 cm.
Waist-Hip Ratio waist circumference | 8 weeks
  The waist-hip ratio will be calculated as an index of body fat distribution. Waist-Hip Ratio will be computed by dividing waist circumference (cm) by hip circumference (cm). Higher Waist-Hip Ratio values will indicate greater central fat accumulation and will be associated with increased cardiometabolic risk.
Walter Reed Visual Assessment Scale | 8 weeks
  self-perception of spinal deformity will be measured using the Walter Reed Visual Assessment Scale. Scores range from 1 to 5, with higher scores indicating greater perceived deformity. Change over 8 weeks will be analyzed.
Scoliosis Research Society-22 Questionnaire Score | 8 weeks
  Quality of life will be assessed using the Scoliosis Research Society-22 questionnaire, which measures function, pain, self-image, mental health, and satisfaction. The total score of the SRS-22 ranges from 22 to 110, with higher scores indicating better quality of life. Total scores will be compared between baseline and 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No